CLINICAL TRIAL: NCT01952912
Title: Comparison of Plasmakinetic Enucleation of the Prostate With Open Prostatectomy for the Treatment of Benign Prostatic Hypertrophy Patients With Large Prostate
Brief Title: Plasmakinetic Enucleation of the Prostate and Open Prostatectomy to Treat Large Prostates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKEP-OP
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2003-12

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PkEP (Active Comparator)
  Interventions: Procedure: PkEP
- OP (Active Comparator)
  Interventions: Procedure: OP

INTERVENTIONS:
Procedure: PkEP
  Arms: PkEP
Procedure: OP
  Arms: OP

SUMMARY:
The investigators hypothesize that Plasmakinetic Enucleation of the Prostate (PkEP) might yield functional results comparable to OP but with lower perioperative morbidity, and have equivalent long-term efficacy with OP for large prostates. The first objective was to demonstrate the non-inferiority of PKEP compared to OP concerning Qmax at one year postoperatively.

To explore the long-term efficacy, we compared the efficacy, safety, and morbidity of PkEP with those of OP in BPH patients with prostate glands larger than 100 g over a follow-up period of 6 years.

ELIGIBILITY:
Inclusion Criteria:

* •Qmax < 12 mL/s, IPSS >19

  * Age between 50 and 70 years
  * Prostate volume larger than 100 mL, as determined by TRUS post-void residual urine volume greater than 50 ml medical therapy failure.

Exclusion Criteria:

* •severe pulmonary disease or heart disease, coagulopathy, neurogenic bladder, bladder calculus, bladder cancer, prostate cancer, urethral stricture and previous prostate or urethral surgery

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-01; Primary Completion 2007-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Qmax at one year postoperatively | 1 year postoperatively

SECONDARY OUTCOMES:
Qmax at other time points after surgery | 1, 3, 6, 24, 36, 48, 60 and 72 months postoperatively
resected adenoma weight | right after the operation
operation time | during the operation
blood loss | perioperatively and on the first postoperative day
postoperative International Prostate Symptom Score | 1, 3, 6, 12, 24, 36, 48, 60 and 72 months postoperatively
duration of catheterization | after the operation
length of postoperative hospital stay | after the operation
QOL | 1, 3, 6, 12, 24, 36, 48, 60 and 72 months postoperatively
PVR | 1, 3, 6, 12, 24, 36, 48, 60 and 72 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Chen S, Zhu L, Cai J, Zheng Z, Ge R, Wu M, Deng Z, Zhou H, Yang S, Wu W, Liao L, Tan J. Plasmakinetic enucleation of the prostate compared with open prostatectomy for prostates larger than 100 grams: a randomized noninferiority controlled trial with long-term results at 6 years. Eur Urol. 2014 Aug;66(2):284-91. doi: 10.1016/j.eururo.2014.01.010. Epub 2014 Jan 24. PMID 24502959